CLINICAL TRIAL: NCT06462547
Title: The ADAPT Study: An Open-label, Long-term Safety Study of INZ-701 in Patients With ENPP1 Deficiency and ABCC6 Deficiency
Brief Title: ADAPT Study: Long-term Safety Study of INZ-701 in Patients With ENPP1 Deficiency and ABCC6 Deficiency
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inozyme Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INZ701-304
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Gene Mutations; Pseudoxanthoma Elasticum; Arterial Calcification; Ectonucleotide Pyrophosphatase/phosphodiesterase1 Deficiency; Autosomal Recessive Hypophosphatemic Rickets Type 2
Keywords: ABCC6; ATP-Binding Cassette Subfamily C Member 6 Deficiency; PXE; Pseudoxanthoma elasticum; GACI; Generalized Arterial Calcification of Infancy; ARHR2; Autosomal Recessive Hypophosphatemic Rickets Type 2; ENPP1; ectonucleotide pyrophosphatase/phosphodiesterase1 deficiency; hypopyrophosphatemia
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Arterial calcification of infancy

STUDY DESIGN:
Intervention Model Description: The ADAPT Study (INZ701-304) is an open-label study to assess the long-term safety of INZ-701 in patients with ENPP1 Deficiency or ABCC6 Deficiency who have received INZ-701 in an existing clinical study and choose to continue dosing for the potential treatment of their condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INZ-701 (Experimental): INZ-701 will be administered by subcutaneous injection on a once-weekly basis as follows:
  * Study participants from 1 year to <13 years of age will receive a dose of 2.4 mg/kg
  * Study participants ≥13 years will either receive a 1.8 mg/kg dose or a 150 mg flat dose of INZ-701
  Interventions: Drug: INZ-701

INTERVENTIONS:
Drug: INZ-701 — INZ-701 is a recombinant fusion protein that contains the extracellular domains of human ENPP1 coupled with an Fc fragment from an immunoglobulin gamma-1 (IgG1) antibody (rhENPP1-Fc).
  Other Names: rhENPP1-Fc

SUMMARY:
The purpose of this study (Study INZ701-304 [ADAPT]) is to assess the long-term safety of INZ-701 in patients with ENPP1 Deficiency or ABCC6 Deficiency who have received INZ-701 in an existing clinical study and choose to continue dosing for the potential treatment of their condition.

DETAILED DESCRIPTION:
The investigational product INZ-701 is being developed as a therapeutic protein for the treatment of ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) Deficiency and adenosine triphosphate (ATP)-binding cassette subfamily C member 6 (ABCC6) Deficiency. INZ-701 is a recombinant fusion protein that contains the extracellular domains of human ENPP1 coupled with an Fc fragment from an immunoglobulin (Ig) G1 antibody.

The ADAPT Study (INZ701-304) is an open-label study to assess the long-term safety of INZ-701 in patients with ENPP1 Deficiency or ABCC6 Deficiency who have received INZ-701 in an existing clinical study and choose to continue dosing for the potential treatment of their condition.

The study will consist of a 30-day Screening Period, followed by an open-label Treatment Period during which all participants will receive once-weekly subcutaneous (SC) doses of INZ-701 and continue with treatment until INZ-701 is commercially available in the country/region of the participant's residence or until Inozyme chooses to discontinue development of INZ-701. Participants will complete an End of Study (EOS) safety follow-up visit approximately 30 days after their last designated study visit assigned by the Investigator and/or Sponsor.

ELIGIBILITY:
Individuals eligible to participate must meet all of the following inclusion criteria:

1. Provide written or electronic informed consent after the nature of the study has been explained, and prior to any research-related procedures, per International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP)
2. Provide assent in accordance with local regulations, if <18 years of age
3. Male or female, greater than 1 year of age
4. Must have completed the protocol-required safety and PK/PD and/or efficacy period(s) of a previous INZ-701 clinical study in ENPP1 or ABCC6 Deficiency, as confirmed by the Sponsor
5. Female participants of childbearing potential who are sexually active must be using or agree to use 1 highly effective form of contraception (per CTFG 2020) from at least 1 month before the first dose of INZ-701 through 30 days after last dose of INZ-701 (greater than 5 half-lives of INZ-701); participants must agree to not donate ova from the period following the first dose of INZ-701 through 30 days after the last dose of INZ-701
6. Male participants who are sexually active must agree to use condoms from the period following the first dose of INZ-701 through 30 days after the last dose of INZ-701; participants must agree to not donate sperm from the period following the first dose of INZ-701 through 30 days after last dose of INZ-701
7. In the opinion of the Investigator, able to complete all aspects of the study

Individuals who meet any of the following exclusion criteria will not be eligible to participate:

1. In the opinion of the Investigator, presence of any clinically significant disease or laboratory abnormality not associated with ENPP1 Deficiency or ABCC6 Deficiency, that will preclude study participation and/or may confound interpretation of study results
2. Known intolerance to INZ-701 or any of its excipients
3. Concurrent participation in another interventional clinical study and/or has received an investigational drug other than INZ-701 within 5 half-lives or within 4 weeks prior to the first dose of INZ-701 in this study, whichever is longer, or use of an investigational device
4. Pregnant, trying to become pregnant, or breastfeeding
5. Male participants trying to father a child

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) | 6 years (long term safety assessment)
  Treatment-emergent AEs are defined as any AE occurring from the first dose of INZ-701 through 30 days after the last dose of INZ-701.
Incidence of Anti-Drug Antibodies (ADA) | 6 years (long term safety assessment)
  For each subject, the presence of ADAs will be assessed and, if present, further evaluation will determine specificity and subtypes.

SECONDARY OUTCOMES:
Time to maximum serum concentration (Tmax) | 6 years (long term safety assessment)
  For each subject, the time to reach maximum concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.
Maximum Plasma Concentration (Cmax) of INZ-701 | 6 years (long term safety assessment)
  For each subject, the maximum concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.collected and assessed.
Mean Change from Baseline in Plasma PPi Concentration | 6 years (long term safety assessment)
  For each subject, their plasma PPi concentrations based on a validated assay will be collected and assessed throughout the study, comparing the participant's baseline value over time.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Gunter, MD, Study Director — Inozyme Pharma, Inc.
Locations (5):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Clinilabs Drug Development Corporation, Eatontown, New Jersey
- Necker-Enfants Malades Hospital, Paris, France
- Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg, Germany
- VCTC, Oxford, United Kingdom